CLINICAL TRIAL: NCT06539143
Title: Analgesia From Conscious Sedation Versus Paracervical Block for Manual Vacuum Aspiration for First Trimester Incomplete Miscarriage in Abakaliki: A Randomized Trial
Brief Title: Analgesia From Conscious Sedation Versus Paracervical Block for Manual Vacuum Aspiration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Darlington-Peter Chibuzor Ugoji (Other)
Responsible Party: Sponsor-Investigator, Darlington-Peter Chibuzor Ugoji, Principal Investigator, Alex Ekwueme Federal University Teaching Hospital
Organization: Alex Ekwueme Federal University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NHREC/16/05/22/209
Record Dates: First submitted 2024-04-14; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Effect of Drug
Keywords: miscarriage; analgesia; manual vacuum aspiration
MeSH Terms: conditions — Abortion, Spontaneous; Agnosia | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: This study is a clinical equivalence randomized controlled trial comparing the efficacy of conscious sedation and paracervical block among women selected for manual vacuum aspiration following incomplete miscarriages in first trimester in Alex Ekwueme Federal University Teaching Hospital, Abakaliki (AEFUTHA), Ebonyi State.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Conscious Sedation) (Active Comparator): 30mg of pentazocine was given intravenously, over one minute and a latency period of about 2 minutes was allowed before starting the procedure for analgesic function to take effect.
  Interventions: Drug: Lidocaine
- GROUP B (The Paracervical Block) (Experimental): Received 10 ml of 1% lidocaine, for the blocks with 4ml at 4 O' clock and 8 O'clock positions and 2 ml at the anterior cervical lip.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — The Paracervical Block with lidocaine for manual vacuum aspiration
  Other Names: Xylocaine

SUMMARY:
Miscarriage is one of the major causes of early pregnancy losses. Incomplete miscarriage is a major cause of maternal morbidity and mortality. Analgesia from both conscious sedation and paracervical could be utilized during manual vacuum aspiration of first trimester incomplete miscarriage. The objectives of this study are to review the existing studies and to compare analgesia from conscious sedation with that of paracervical block among women selected for manual vacuum aspiration following first trimester incomplete miscarriages in Alex Ekwueme Federal University Teaching Hospital, Abakaliki [AEFUTHA].

DETAILED DESCRIPTION:
SUMMARY

Background:

First trimester pregnancy losses are estimated to occur in 14-19% of all clinically confirmed pregnancies and account for about 80% of all the pregnancy losses. Miscarriage is one of the major causes of early pregnancy losses. Incomplete miscarriage is a major cause of maternal morbidity and mortality.

Analgesia from both conscious sedation and paracervical could be utilized during manual vacuum aspiration of first trimester incomplete miscarriage. In my center, conscious sedation is mostly used but because of the pronounced systemic side effect of drowsiness, weakness etc, there is a shift to paracervical block hence this study.

Objectives:

The objectives of this study are to review the existing studies and to compare analgesia from conscious sedation with that of paracervical block among women selected for manual vacuum aspiration following first trimester incomplete miscarriages in Alex Ekwueme Federal University Teaching Hospital, Abakaliki [AEFUTHA].

Methodology:

This was a randomized control trial equivalent study that compared the analgesia from conscious sedation with that of the paracervical block in women selected for manual vacuum aspiration following first trimester incomplete miscarriage in AEFUTHA. Patients were categorized into groups: A and B. Those in group A received conscious sedation using intravenous diazepam 10 mg and intravenous pentazocine 30 mg stat while those in the other group B received paracervical block via the use of 10ml of 1% lidocaine with 4ml at 4:00 clock and 8:00 clock respectively and 2ml at the anterior lip of the cervix. After analgesic effect has occurred, manual vacuum aspiration was done and there after pain assessment was be carried out at 10 mins, 2 hours, 6 hours, 12 hours and 24 hours respectively. The vital signs and oxygen saturation pre and post operatively were monitored with chart kept for analysis.

Analysis:

The data were analyzed using Spss, version 28.0 (2022). Continuous variables were compared with t- test while categorical variables were compared with Chi- square and the p-value determined. P- value less than 0.05 was taken to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* - Between the ages of 18- 45 years.
* Spontaneous incomplete miscarriage at less than 13 weeks.
* Not allergic to drugs for the study
* Patients that give consent

Exclusion Criteria:

* - Patients who do not consent to MVA [ Manual vacuum aspiration].
* Those with known allergy history to the drug agents.
* Those with septic incomplete miscarriage.
* Patients with infection at the cervical blocking sites.
* Those with active pelvic inflammatory disease.
* Patients with neurological or psychiatric disease.
* Incomplete miscarriage at greater than 13 weeks.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This is by physical examination
Enrollment: 81 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Mean pain score using the Visual analogue scale | Pain and side effects experienced following the use of the analgesic agents at about 10 minutes, 2 hours, 6 hours, 12 hours and 24 hours following the procedure was noted. Higher score showed more pain and lower score showed lower pain
  The primary outcome measure is the mean pain score of the participants in the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: DARLINTON-PETER CHIBUZOR C UGOJI, MBBS, Principal Investigator — Alex Ekwueme Federal University Teaching Hospital
Locations (1):
- AEFUTHA, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No
This will only be after full defense of the work at the college

REFERENCES:
- [Background] Sotiriadis A, Makrydimas G, Papatheodorou S, Ioannidis JP. Expectant, medical, or surgical management of first-trimester miscarriage: a meta-analysis. Obstet Gynecol. 2005 May;105(5 Pt 1):1104-13. doi: 10.1097/01.AOG.0000158857.44046.a4. PMID 15863551